CLINICAL TRIAL: NCT00499434
Title: Correlation Between Values of Serum Cytokines and of Those Dosed by mRNA Expression Through the Use of Real-time PCR and Hepatic Histology in Patients Infected by HIV-1 and the Hepatitis-C Virus
Brief Title: Correlation Between Cytokines and Hepatic Histology in Patients Infected by HIV-1 and the Hepatitis-C Virus
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: Alexandre Naime Barbosa, SAE e Hospital Dia de Aids - Faculdade de Medicina de Botucatu - Unesp
Other Study IDs: upeclin/HC/FMB-Unesp-14
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Last update posted 2009-12-04 (Estimated); Status verified 2009-12

CONDITIONS: Acquired Immune Deficiency Syndrome; Hepatitis, Viral, Non-A, Non-B, Parenterally-Transmitted; HIV Infections
Keywords: aids
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hepatitis C; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study aims at correlating TNF-α, INF-γ, IL-2, IL-4, IL-10 and TGF-β values as dosed by ELISA and mRNA expression by real-time PCR with histopathological hepatic biopsy findings in individuals with HIV/HCV coinfection. This population will be divided into three groups (G1: with no HAART; G2: with detected HIV viral load (HIV VL); G3: with undetected HIV VL), which will be then compared to two control groups with monoinfection by HIV or by HCV, in addition to a third control group comprising normal blood donors.

DETAILED DESCRIPTION:
Infection by the hepatitis-C virus (HCV) in people living with HIV/AIDS (PLHA) has progressively gained distinction since the survival increase generated by the use of highly active antiretroviral therapy (HAART) has enabled the presentation of complications from HCV chronic infection. There are approximately 10 million coinfected individuals, that is, 25% of the total PLHA as both viruses share transmission routes.

HCV infection can be regarded as an opportunistic disease in this population once there is the acceleration of its natural history represented by the HCV high viral load, early hepatic fibrosis and greater occurrence of steatosis, cirrhosis and hepatocellular carcinoma, leading to greater morbid-mortality by terminal hepatic disease. The scenario is not also favorable as regards HCV treatment, since the response rate in coinfected individuals is significantly lower than in mono-infected HCV patients.

The complex relationship between immune response and HCV determines the velocity and the distinct outcomes found. The major determinant for the development of cirrhosis and hepatic insufficiency is the accumulation of fibrosis and inflammatory activity closely related to collagen synthesis by fibroblasts and hepatocyte-apoptosis induction related to TGF-β production. In individuals with more severe hepatic lesion, there is the prevalence of expression of the Th-2 profile in the peripheral blood, which is characterized by high levels of IL-4 and IL-10, whereas, in the hepatic tissue, a larger expression of cytokines of the Th-1 profile, such as IL-2 and INF-γ, is observed. This phenomenon is known as "compartmentalization" of the immune response.

If the immunopathogenic dynamics is already complex in HCV mono-infected individuals, in the HIV/HCV coinfection condition, few studies specifically approach the topic, without, however, evaluating the correlation between specific T-cell response and hepatic-lesion staging. In HIV mono-infected patients without antiretroviral treatment and with disease progression, the prevalence of the Th-0/Th-2 profile is observed, which is particularly influenced by IL-10 increase. Even in individuals treated by HAART, there is no recovery of the capacity to express the Th-1 profile, and most of such patients show the mature Th-0 profile and low IL-2 levels.

HCV viral load in PLHA is higher in both the plasma and the hepatic tissue, and the replication of HCV in macrophages, CD4 and CD8 T lymphocytes as well as in lymphnodes is also observed in such condition. TGF-β is particularly high in this coinfection, thus justifying the onset of faster fibrosis. The reduction of CD8 T lymphocyte response to IFN-γ also occurs, which favors the persistence of infection and prevents specific T-cell response. As regards HIV treatment, there is evidence that coinfected patients non-treated by HAART tend to present a Th-2 profile more often than treated individuals, without, however, significant differences in TGF-β levels.

Due to the lack of studies correlating the production tendencies of both pro-inflammatory and fibrogenesis-inducing cytokines with histopathological findings from hepatic biopsy in coinfected individuals, investigations are necessary in order establish parameters that will allow the prediction of a better or worse prognosis and also more accurately indicate the performance of hepatic biopsy.

This study aims at correlating TNF-α, INF-γ, IL-2, IL-4, IL-10 and TGF-β values as dosed by ELISA and mRNA expression by real-time PCR with histopathological hepatic biopsy findings in individuals with HIV/HCV coinfection. This population will be divided into three groups (G1: with no HAART; G2: with detected HIV viral load (HIV VL); G3: with undetected HIV VL), which will be then compared to two control groups with monoinfection by HIV or by HCV, in addition to a third control group comprising normal blood donors.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HIV infection or aids
* Diagnosis of chronic hepatitis C

Exclusion Criteria:

* Other hepatic diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: SAE e Hospital Dia de Aids patients
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2007-08; Primary Completion 2009-01 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
This study aims at correlating TNF-α, INF-γ, IL-2, IL-4, IL-10 and TGF-β values as dosed by ELISA and mRNA expression by real-time PCR with histopathological hepatic biopsy findings in individuals with HIV/HCV coinfection | Two years

SECONDARY OUTCOMES:
This study aims at correlating TNF-α, INF-γ, IL-2, IL-4, IL-10 and TGF-β values as dosed by ELISA and mRNA expression by real-time PCR with CD4 and HIV viremia values in individuals with HIV/HCV coinfection | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre N Barbosa, MD, MSc, Principal Investigator — UPECLIN HC FM Botucatu Unesp
Locations (1):
- SAE e Hospital Dia de Aids, Botucatu, São Paulo, Brazil